CLINICAL TRIAL: NCT04994340
Title: Physical Activity Observatory of Castilla-La Mancha
Acronym: OBAFIT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Castilla-La Mancha (Other)
Collaborators: Consejería de Educación, Cultura y Deportes de Castilla-La Mancha (Unknown); Dirección General de Juventud y Deportes de Castilla-La Mancha (Unknown)
Responsible Party: Principal Investigator, Javier Valenciano, Principal Investigator, University of Castilla-La Mancha
Other Study IDs: 2020/01/007
Record Dates: First submitted 2021-07-28; First posted 2021-08-06 (Actual); Last update posted 2021-08-06 (Actual); Status verified 2021-08

CONDITIONS: Sedentary Behavior; Exercise; Physical Fitness
Keywords: Childhood; Physical activity; Health; School; Surveillance
MeSH Terms: conditions — Sedentary Behavior; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Children: From a cross-sectional perspective, children will fill out questionnaires related to their subjective physical activity levels (PAQ-C), levels of sedentary activity (YLSBQ), and socio-economic status (Family Affluence Scale III) during school hours. Two sessions of physical education will be used to measure the health-related physical fitness of children through the ALPHA-Fitness battery test. The sequence to administer this battery will be: 1. Weight and height (BMI); 2. Waist circumference; 3. Skin folds; 4. Hand grip strength, long jump with feet together, and 4x10 m shuttle run test (these tests could be carried out alternately or simultaneously since there will always be 2 or more evaluators); 5. 20 m Course Navette test.
- Adolescents: From a cross-sectional perspective, adolescents will fill out questionnaires related to their subjective physical activity levels (PAQ-A), levels of sedentary activity (YLSBQ), and socio-economic status (Family Affluence Scale III) during school hours. Two sessions of physical education will be used to measure the health-related physical fitness of adolescents through the ALPHA-Fitness battery test. The sequence to administer this battery will be: 1. Weight and height (BMI); 2. Waist circumference; 3. Skin folds; 4. Hand grip strength, long jump with feet together, and 4x10 m shuttle run test (these tests could be carried out alternately or simultaneously since there will always be 2 or more evaluators); 5. 20 m Course Navette test.

SUMMARY:
The OBAFIT project aims to examine the patterns of physical activity, sedentary activity and health-related physical fitness of the boys and girls enrolled in schools of Primary Education and Secondary Education in Castilla-La Mancha (Spain). The design of the project is observational/cross-sectional. Through an epidemiological orientation, it proposes a representative sampling of a multistage type of the Castilian-La Mancha population aged 6 to 16 years. The subjects that will make up the sample will be selected from among the 724 Castilian-La Mancha schools with teachings in the Primary Education stage, and among 373 Secondary Education schools. To ensure the heterogeneity of the population, both public and private centers will be selected, and proportionally between centers that have Healthy School Programs (PES) from those that do not. The sample will be multistage, randomized and stratified according to province (Albacete, Ciudad Real, Cuenca, Guadalajara and Toledo), area (urban, semi-urban, rural), sex (men, women) and age (one group for each age group).

DETAILED DESCRIPTION:
The OBAFIT project was designed to provide a public tool where PA habits, sedentary behaviors and the health-related physical fitness of school children from Castilla-La Mancha (a Spanish region) could be visualized. OBAFIT also allows physical education teachers at participating schools to monitor and observe the evolution of these variables in their students.

For this, the schooling data provided by the Consejería de Educación, Cultura y Deportes de la Junta de Comunidades de Castilla-La Mancha (Ministry of Education, Culture and Sports of the Community Board of Castilla-La Mancha) are considered: the population enrolled in the region from the first to the sixth year of Primary Education amounts to 131,903 students (63,488 girls; 68,415 boys) distributed in the five provinces (Albacete 24,143; Ciudad Real 31,053; Cuenca 11,001; Guadalajara 17,560; Toledo 48,146) both in public (106,366) and private (25,537) schools.

In the case of Secondary Education and the first year of high school, the number of students stands at 98,745 (50,807 men and 49,267 women) from the five provinces of the region (Albacete 19,016; Ciudad Real 23,599; Cuenca 8,971; Guadalajara 12,827; Toledo 34,332) of public centers (80,996) and private (19,078).

The sample size, calculated through the Edidat 4.2 software, is 631 subjects for the Primary sample and 631 for the Secondary sample (assuming normal distribution). A confidence level of 95% and a margin of error of 3% have been considered, and the CVR associated with low CRC with a prevalence of 18% is assumed as the parameter of greater variance. If the same level of confidence and margin of error for both sexes are considered, the sample would amount to 1,262 for each educational level. Assuming a non-response rate of 30%, the final sample size is estimated at 1640 students in Primary Education and 1640 for Secondary Education.

The participants that will make up the sample will be selected from the 724 Castilian-La Mancha schools with education in the Primary Education stage, and from 373 Secondary Education centers. Both public and private centers will be selected. The sample will be multistage, randomized and stratified according to province (Albacete, Ciudad Real, Cuenca, Guadalajara and Toledo), area (urban, semi-urban, rural), gender (men, women) and age (one group for each section of age).

Once the sample size has been determined, a lottery of schools classified based on the aforementioned criteria is carried out, considering in all cases the proportionality in the number of students. For this, a multistage method with proportional probability will be used using SPSS 24.0 software. Approximately 48 centers for Primary Education and 55 for Secondary Education will be selected, taking into account that there are 6 Primary courses and 4 in E.S.O. (Spanish system) in addition to 1st year of high school In the selected schools, three boys and three girls will be randomly chosen per group-class and level, on which the different instruments will be applied. A priori, due to pedagogical and operational issues in the administration, proportional age preselection will not be carried out (for the same group-class). Since all students in the same class-group will have the same probability of being selected, the age and sex quotas will be corrected at the end of data collection by a weighting system.

ELIGIBILITY:
Inclusion Criteria:

- Be enrolled in any school in Castilla-La Mancha (primary or secondary, public or private, rural or urban).

Exclusion Criteria:

* Temporary injury or disability that prevents physical testing.
* Clinical diagnosis of diabetes or diseases not related to nutrition.

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Boys and girls aged 6 to 16 years enrolled in Primary and Secondary Education schools in Castilla La Mancha.
Sampling Method: Probability Sample
Enrollment: 3280 (Estimated)
Dates: Start 2017-09-08 (Actual); Primary Completion 2018-06-23 (Actual); Study Completion 2022-06-23 (Estimated)

PRIMARY OUTCOMES:
Subjective physical activity levels | 2017/2018 to 2021/2022
  Physical activity assessed by self-report (PAQ-C or PAQ-A). The scales ranged from 0 to 5, where higher values indicate greater levels of physical activity.
Device-measured physical activity levels | 2017/2018 to 2021/2022
  Physical activity assessed by accelerometer (Measure carried out only in those schools that give consent)
Sedentary behavior | 2017/2018 to 2021/2022
  Sedentary behavior assessed by self-report (YLSBQ)
Sedentary behavior | 2017/2018 to 2021/2022
  Adolescents' sedentary behaviors assessed by self-report (ASAQ)
Health-related physical fitness | 2017/2018 to 2021/2022
  Health-related physical fitness assessed by the ALPHA-FITNESS test battery

SECONDARY OUTCOMES:
Socioeconomic status | 2017/2018 to 2021/2022
  Socioeconomic status assessed by the Family Affluence Scale III. The scale ranged from 0 to 13, where higher values indicate a greater socioeconomic status.

OTHER OUTCOMES:
Age | 2017/2018 to 2021/2022
  Age assessed by self-report
Gender | 2017/2018 to 2021/2022
  Gender assessed by self-report
Body mass index | 2017/2018 to 2021/2022
  Body mass calculated through height and weight measurements
Type of school | 2017/2018 to 2021/2022
  Public/private schools or urban/semirural/rural schools extracted from the registry of Castilla-La Mancha

CONTACTS AND LOCATIONS:
Overall Officials: Javier Valenciano, PhD, Principal Investigator — University of Castilla-La Mancha; Juan Gregorio Fernández-Bustos, PhD, Principal Investigator — University of Castilla-La Mancha
Locations (1):
- Universidad Castilla-La Mancha, Toledo, Spain

REFERENCES:
- [Background] Poitras VJ, Gray CE, Borghese MM, Carson V, Chaput JP, Janssen I, Katzmarzyk PT, Pate RR, Connor Gorber S, Kho ME, Sampson M, Tremblay MS. Systematic review of the relationships between objectively measured physical activity and health indicators in school-aged children and youth. Appl Physiol Nutr Metab. 2016 Jun;41(6 Suppl 3):S197-239. doi: 10.1139/apnm-2015-0663. PMID 27306431
- [Background] Biddle SJ, Gorely T, Pearson N, Bull FC. An assessment of self-reported physical activity instruments in young people for population surveillance: Project ALPHA. Int J Behav Nutr Phys Act. 2011 Jan 2;8:1. doi: 10.1186/1479-5868-8-1. PMID 21194492
- [Background] Benitez-Porres J, Lopez-Fernandez I, Raya JF, Alvarez Carnero S, Alvero-Cruz JR, Alvarez Carnero E. Reliability and Validity of the PAQ-C Questionnaire to Assess Physical Activity in Children. J Sch Health. 2016 Sep;86(9):677-85. doi: 10.1111/josh.12418. PMID 27492937
- [Background] Cain KL, Sallis JF, Conway TL, Van Dyck D, Calhoon L. Using accelerometers in youth physical activity studies: a review of methods. J Phys Act Health. 2013 Mar;10(3):437-50. doi: 10.1123/jpah.10.3.437. PMID 23620392
- [Background] Hidding LM, Chinapaw MJM, van Poppel MNM, Mokkink LB, Altenburg TM. An Updated Systematic Review of Childhood Physical Activity Questionnaires. Sports Med. 2018 Dec;48(12):2797-2842. doi: 10.1007/s40279-018-0987-0. PMID 30298479
- [Background] Ortega FB, Ruiz JR, Castillo MJ, Moreno LA, Gonzalez-Gross M, Warnberg J, Gutierrez A; Grupo AVENA. [Low level of physical fitness in Spanish adolescents. Relevance for future cardiovascular health (AVENA study)]. Rev Esp Cardiol. 2005 Aug;58(8):898-909. Spanish. PMID 16053823
- [Background] Ruiz JR, Espana Romero V, Castro Pinero J, Artero EG, Ortega FB, Cuenca Garcia M, Jimenez Pavon D, Chillon P, Girela Rejon MJ, Mora J, Gutierrez A, Suni J, Sjostrom M, Castillo MJ. [ALPHA-fitness test battery: health-related field-based fitness tests assessment in children and adolescents]. Nutr Hosp. 2011 Nov-Dec;26(6):1210-4. doi: 10.1590/S0212-16112011000600003. Spanish. PMID 22411362
- [Background] Marasso D, Lupo C, Collura S, Rainoldi A, Brustio PR. Subjective versus Objective Measure of Physical Activity: A Systematic Review and Meta-Analysis of the Convergent Validity of the Physical Activity Questionnaire for Children (PAQ-C). Int J Environ Res Public Health. 2021 Mar 25;18(7):3413. doi: 10.3390/ijerph18073413. PMID 33806106
- See also: OBAFIT website — https://obafi.es/